CLINICAL TRIAL: NCT04549038
Title: Time Restricted Nutrition in Pediatric Stem Cell Transplant Recipients: Impact on Circadian Rhythm, Insulin Regulation, and Outcomes
Brief Title: Time Restricted Nutrition in Pediatric Stem Cell Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-1180
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Hematopoietic Stem Cell Transplant
MeSH Terms: interventions — Nutritional Status

STUDY DESIGN:
Intervention Model Description: 1:1 randomized, non-blinded, controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cases (Experimental): Patients randomized to the cases group will receive their nutrition over a period of 12-16 hours, with minimum 8 hours of fasting and maximum 12 hours of fasting. All patients will receive 100% of their daily nutrition.
  Interventions: Other: 12-16 hour nutrition
- Controls (No Intervention): Patients randomized to the control group will receive the current standard of care (24-hour continuous nutrition). All patients will receive 100% of their daily nutrition.

INTERVENTIONS:
Other: 12-16 hour nutrition — Cases will receive their nutrition over a period of 12-16 hours, with minimum 8 hours of fasting and maximum 12 hours of fasting. Feeding will begin in morning hours unless otherwise directed by an investigator or registered dietician.
  Arms: Cases

SUMMARY:
Circadian cycles, metabolism, and nutrition are intimately linked, and the timing of meals play an important role in synchronizing peripheral circadian rhythms. There are little data describing the influence of nocturnal feeds on sleep, metabolism, and overall health in hospitalized children. To evaluate this association, the investigators will conduct a single-center, randomized, non-blinded controlled trial that will test the impact of nocturnal enteral/parenteral nutrition on patient outcomes.

DETAILED DESCRIPTION:
HSCT provides a potential cure for children and adults with high risk and relapsed malignancy, immune deficiency, and other fatal illnesses. Circadian cycles, metabolism, and nutrition are intimately linked, and the timing of meals play an important role in synchronizing peripheral circadian rhythms; however, the standard of care for HSCT recipients is to deliver continuous feeds (either enterally or parenterally).

The objective of this study is to evaluate the influence of the timing of feeding on sleep and metabolism in HSCT subjects. The investigators hypothesize patients receiving feeds during daytime hours (0800-2000) in comparison to continuous (24 hours), will have improved sleep efficiency, decreased blood glucose, insulin, and triglycerides over patients who receive feeding overnight. The aim of this study is to evaluate the influence of the timing of feeds on sleep, metabolism, and outcomes in HSCT subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients >/= 12 months of age undergoing HSCT and receiving a myeloablative preparative regimen

Exclusion Criteria:

* Prior history of hypoglycemia, diabetes mellitus, metabolic disease, or other requirement for continuous nutrition

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-05-19 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
Number of wake episodes | 21 days
  Number of wake episodes
Duration of wake episodes | 21 days
  Duration of wake episodes

SECONDARY OUTCOMES:
Hypertension | 21 days
  Incidence of hypertension
Weight change | 21 days
  Change in weight at day +7, +14, and +21 from day 0
Time to tolerating oral feeds | 21 days
  Number of days post-transplant until the patient tolerates feeds/nutrition
Neutrophil engraftment | 21 days
  Time to absolute neutrophil count >500
Cortisol levels | 21 days
  3 times weekly morning cortisol levels
Triglyceride levels | 21 days
  Weekly triglyceride levels
Glucose levels | 21 days
  Daily glucose levels

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Dandoy, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No